CLINICAL TRIAL: NCT04703673
Title: Non-interventional Study on the Quality of Life Before and After Intake of Sinolpan® (Forte) in Inflammatory Diseases of the Respiratory Tract - an Anonymous Patient Survey
Brief Title: Sinolpan® Pharmacy Non-interventional Study - Quality of Live
Status: Completed | Type: Observational
Sponsor: Engelhard Arzneimittel GmbH & Co.KG (Industry)
Collaborators: ClinCompetence Cologne GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: EA-20-01-996
Record Dates: First submitted 2020-12-17; First posted 2021-01-11 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Rhinosinusitis Acute; Rhinosinusitis Chronic; Bronchitis
Keywords: Quality of Life
MeSH Terms: conditions — Bronchitis | interventions — Eucalyptol; Nasal Decongestants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sinolpan® group: Sinolpan® group: patients suffering from rhinosinusitis and, where appropriate, from bronchitis; intake of Sinolpan® 100 mg or Sinolpan® forte 200 mg (cineol) according to the instructions for use; before and after treatment for rhinosinusitis and, where appropriate, from bronchitis, patients complete a questionnaire that contains the Rhinosinusitis Quality of Life questionnaire and Questions about the severity of bronchitis symptoms. The latter should only be answered by patients who suffer from bronchitis in addition to rhinosinusitis.
  Interventions: Drug: Cineole
- Nasal spray group: Control group: patients with rhinosinusitis; Use of nasal decongestants according to the instructions for use. Before and after treatment for rhinosinusitis, patients complete a questionnaire that includes the Rhinosinusitis Quality of Life questionnaire.
  Interventions: Drug: Nasal Decongestant

INTERVENTIONS:
Drug: Cineole — self administration according to directions for use
  Groups: Sinolpan® group
Drug: Nasal Decongestant — self administration according to directions for use
  Other Names: nasally applied α-sympathomimetics
  Groups: Nasal spray group

SUMMARY:
This non-interventional study investigates the Quality of Life of patients suffering from rhinosinusitis. Patients who seek advice in a pharmacy and choose to intake Sinolpan® or Sinolpan® forte or to use nasally applied α-sympathomimetics can participate in this anonymous patient survey.

DETAILED DESCRIPTION:
Within the scope of this non-interventional observational study, the quality of life of rhinosinusitis patients under self-medication with the 1,8 - cineole preparation Sinolpan® or Sinolpan® forte (Sinolpan® group) or with a nasally applied α-sympathomimetic (control group) is investigated during conditions of daily life. Patients who seek advice from a pharmacy regarding the treatment of their symptoms and who choose Sinolpan® (forte) or a nasal α-sympathomimetic can participate in this study and are asked to complete a questionnaire before and after the treatment. For organizational reasons, the recruitment of patients for the Sinolpan® group (planned number of patients: 500) or the control group (planned number of patients: 50) is conducted in different pharmacies.

The primary objective of this anonymous data collection is to assess the quality of life in patients with rhinosinusitis. The German version of the Rhinosinusitis Quality of Life questionnaire, which was only recently validated in a doctoral thesis, is used for this purpose. Additionally, for patients in the Sinolpan® group who also suffer from bronchitis, the bronchitis severity score is determined. In addition, data on side effects and tolerability of the treatment as well as on patients' satisfaction are collected.

ELIGIBILITY:
Inclusion Criteria:

* Suitable patients for the Sinolpan® group are patients aged 18 years or older who seek advice from a pharmacy regarding the treatment of their acute or chronic (rhino) sinusitis and, where appropriate, their bronchitis and who choose the intake of Sinolpan® (forte) for therapy.
* Suitable patients for the control group are patients aged 18 years or older who seek advice from a pharmacy regarding the treatment of their acute or chronic (rhino) sinusitis and who choose to apply nasal α-sympathomimetics for therapy.

Exclusion Criteria:

* According to the instructions for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory diseases of the respiratory tract
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the Rhinosinusitis Quality of Life Score | Baseline (before first administration) and at day 10 resp. after end of treatment
  The Rhinosinusitis Quality of Life is a validated questionnaire (Atlas et al., Qual Life Res 2005, 14, 1375-1386). It includes 5 symptom severity items (sinus headache/facial pain/facial pressure, blocked or stuffy nose, post-nasal drip, thick nasal discharge, runny nose).
  It also includes 9 symptom impact items (tired or fatigued, trouble sleeping, harder to concentrate, harder to do the things you normally do, embarrassed, frustrated, irritable, sad or depressed, think about).
  The score of the frequency of severity items and the score of the symptom impact items covers a Likert-scale: 1 to 5 with 1 = none of the time, 2= a little of the time, 3 = some of the time, 4 = most of the time and 5 = all of the time.
  The score of the bothersomeness covers a scale from (not bothered at all) to 10 (bothered a lot).
  The sum values of the individual subscores are normalised towards 100, resulting in values between 0 and 100.

SECONDARY OUTCOMES:
Bronchitis severity score (BSS) | Baseline (before first administration) and at day 10 resp. after end of treatment
  For patients suffering additionally from bronchitis: severity of bronchitis Symptoms
  The BSS comprises the following five symptoms typical for acute bronchitis:
  cough, sputum, rales on auscultation, chest pain on coughing, and dyspnoea. These symptoms are each assessed according to a 5-point Likert scale: 0=absent, 1=mild, 2=moderate, 3=severe and 4=very severe. The points allocated to each of the symptoms are added to make the total score. This can therefore vary between 0 and 20 points and should show a one-dimensional degree of severity in the clinical signs of acute bronchitis.
Number of adverse drug reactions | During the treatment period (maximum of 10 days)
  Number of adverse drug reactions, the reported nature of ADR, the duration and the incidence of ADRs
Tolerability of the Treatment score | Query on the last day of treatment (maximum day 10)
  Tolerability will be assessed by the participants by means of the following 4-point-tolerability score: very good, good, satisfactory, not satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Prof, Study Director — ClinCompetence Cologne GmbH
Locations (1):
- ClinCompetence Cologne GmbH, Cologne, Germany